CLINICAL TRIAL: NCT02895906
Title: A 5-Week, Multi-center, Open-label Study to Assess the Safety and Efficacy of NFC-1 in Subjects Aged 12-17 Years With 22q11.2 Deletion Syndrome and Commonly Associated Neuropsychiatric Conditions (Anxiety, ADHD, ASD)
Brief Title: Safety and Efficacy Study of NFC-1 in Subjects Aged 12-17 Years With 22q11.2DS & Associated Neuropsychiatric Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDGN-NFC1-22Q-101
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: 22q11.2 Deletion Syndrome
Keywords: 22q11.2 DS
MeSH Terms: conditions — DiGeorge Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NFC-1 (Experimental): Doses of NFC-1 will be administered as 50, 100, 200, or 400 mg twice daily as capsules for oral administration.
  Interventions: Drug: NFC-1

INTERVENTIONS:
Drug: NFC-1 — Doses of NFC-1 will be administered as 50, 100, 200, or 400 mg twice daily as size 2, hard gelatin capsules for oral administration.
  Other Names: NFC1

SUMMARY:
This is a 5-week, multi-center, open-label, dose optimization trial in subjects aged 12-17 years with 22q11DS who have a diagnosis of anxiety disorder, and/or ADHD, and/or ASD. Approximately 12 subjects will be initiated, dose optimized, and maintained on NFC-1 over a period of 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of a 22q11.2 deletion prior to screening.
* Subject has a diagnosis of anxiety disorder and/or ADHD and/or ASD based upon diagnostic evaluations performed at screening, history, and clinical judgement.
* Subject is judged to be in general good health, other than having anxiety disorder and/or ADHD and/or ASD and 22q11DS. Medical conditions related to 22q11DS must be clinically stable post surgical correction and/or medical management.
* Subject has no clinically significant abnormality on 12-lead electrocardiogram (ECG) performed at screening or baseline such as serious arrhythmia, bradycardia, tachycardia, cardiac conduction problems, or other abnormalities deemed to be a potential safety issue.
* Subject and parent/legal guardian understand the study procedures and agree to the subject's participation in the study as indicated by parental/legal guardian signature on the subject informed consent form and subject's signature on the assent form.

Exclusion Criteria:

* Subject has a diagnosis of co-morbid major psychiatric disorders (ie, aside from anxiety disorder, ADHD, and/or ASD), including major depression, bipolar disease, schizophrenia (or any psychotic disorder), and moderate or severe intellectual disability, which in the opinion of the investigator may interfere with the conduct of study evaluations.
* Subject has an IQ < 65 as determined by the Wechsler Abbreviated Scale of Intelligence.
* Subject has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject by his/her participation in the study.
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or disease which is not currently stable clinically. Subjects with a history of uncomplicated kidney stones may be enrolled in the study at the discretion of the investigator.
* Subject has a history of stroke, chronic seizures, or other major neurological disorder which, in the opinion of the investigator, would interfere with the subject's ability to participate and/or be evaluated in the trial.
* Subject is currently considered at risk for suicide (in the opinion of the investigator), has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.
* Subject has taken any antidepressants, antipsychotics, anxiolytics, or non-stimulant ADHD medication within 30 days of the Screening Visit.
* Subject is taking a prohibited medication

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Time to symptom relapse | Through study completion, up to 5 weeks

SECONDARY OUTCOMES:
Response to treatment based on Clinical Global Impression - Improvement scale | Through study completion, up to 5 weeks
Safety and tolerability as determined by AEs, laboratory results, C-SSRS, and K-SADS | Through study completion, up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glessner JT, Khan ME, Chang X, Liu Y, Otieno FG, Lemma M, Slaby I, Hain H, Mentch F, Li J, Kao C, Sleiman PMA, March ME, Connolly J, Hakonarson H. Rare recurrent copy number variations in metabotropic glutamate receptor interacting genes in children with neurodevelopmental disorders. J Neurodev Disord. 2023 Apr 29;15(1):14. doi: 10.1186/s11689-023-09483-z. PMID 37120522
- [Derived] Slaby I, Hain HS, Abrams D, Mentch FD, Glessner JT, Sleiman PMA, Hakonarson H. An electronic health record (EHR) phenotype algorithm to identify patients with attention deficit hyperactivity disorders (ADHD) and psychiatric comorbidities. J Neurodev Disord. 2022 Jun 11;14(1):37. doi: 10.1186/s11689-022-09447-9. PMID 35690720